CLINICAL TRIAL: NCT01316952
Title: A Nested Case-control Study of the Association Between Coreg IR and Coreg CR and Hypersensitivity Reactions: Anaphylactic Reaction/Angioedema-Updated Analysis
Brief Title: Coreg and HSRs-Updated Analysis
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114522; WEUSRTP4862 (Other: GSK)
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Hypersensitivity
Keywords: carvedilol; propranolol; hypersensitivity reactions; beta- blockers; Coreg
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LabRx database Oct. 1st 2004 to Sep. 30th 2009: The study cohort from which cases and controls are drawn is all subjects in the LabRx database between Oct. 1st 2004 to Sep. 30th 2009.
  Interventions: Drug: Carvedilol immediate release only; Drug: Carvedilol extended release only; Drug: Long acting β-blockers; Drug: Other α1/β-adrenergic antagonists; Drug: Short acting Non-selective β-blockers and short acting β1-Selective agents; Other: No β-blocker

INTERVENTIONS:
Drug: Carvedilol immediate release only — All dosages of carvedilol immediate release
Drug: Carvedilol extended release only — All dosages of carvedilol extended release
Drug: Long acting β-blockers — All dosages of LA propranolol and SA metoprolol
Drug: Other α1/β-adrenergic antagonists — i.e., labetalol. All dosages. Excluding carvedilol immediate release and carvedilol extended release.
Drug: Short acting Non-selective β-blockers and short acting β1-Selective agents — All dosages of short acting non-selective β-Blockers (Carteolol, Levobunolol, Metipranolol, Nadolol, Penbutolol, Pindolol, Sotalol, Timolol) and short acting β1-Selective agents (Acebutolol, Atenolol, Betaxolol, Bisoprolol, Nebivolol)
Other: No β-blocker — No β-blocker within the month prior to the index date

SUMMARY:
A cluster of reports of hypersensitivity reactions among patients who switched from carvedilol (immediate release formulation, referred to hereafter as carvedilol) to carvedilol extended release was received during the initial post-launch period of carvedilol extended release. In follow up to this observation, product labeling for both agents was updated and a nested case control study was subsequently conducted to examine the risk of serious hypersensitivity reactions i.e. anaphylactic reaction and/or angioedema among patients who used carvedilol extended release compared to carvedilol and separately compared to other long acting beta(β)-blockers. This proposed analysis is an update to the previously conducted analysis using the same database, LabRx, now containing 2 additional years of data, which should provide a larger number of carvedilol extended release exposed subjects.

ELIGIBILITY:
Inclusion Criteria:

* At least one prescription claim for a β-blocker during follow-up time available in the database.
* At least one month of enrollment in the healthcare plan

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Derived from the LabRx database from Oct. 1st 2004 to Sep. 30th 2009. The LabRx Database (referred to in publications as the "i3 InVision Data Mart") is provided by Ingenix Pharmaceutical Services, Inc. It is a comprehensive, de-identified U.S. healthcare claims database that contains the aggregated health claims experience of the covered lives managed by United Healthcare. It contains only those covered lives for which there exists a combined benefit structure including medical and prescription coverage. Overall, it is representative of the non-elderly, insurance-carrying population in the U.S., but it also contains information on several hundred thousand Managed Medicaid and Medicare Advantage members. It contains inpatient, outpatient and pharmacy claims, lab results and enrolment information on over 30.5 million lives from October 2004 through September 2009.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Hypersensitivity reactions (anaphylactic reaction/ angioedema) | Hypersensitivity reactions among users in the LabRx database between Oct. 1st 2004 to Sep. 30th 2009

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Koro CE, Sowell MD, Stender M. An assessment of the association between carvedilol exposure and severe hypersensitivity reactions, angioedema, and anaphylactic reactions: a retrospective nested case-control analysis. Clin Ther. 2012 Apr;34(4):870-7. doi: 10.1016/j.clinthera.2012.02.027. Epub 2012 Mar 22. PMID 22444788